CLINICAL TRIAL: NCT06920732
Title: Comparative Efficacy of 3L and 2L Integrated Techniques for Gynecologic Cancer-related Lower Extremity Lymphedema: a Retrospective Study
Status: Completed | Type: Observational
Sponsor: Zunyi Medical College (Other)
Responsible Party: Principal Investigator, Deng Chengliang, Director of the Department of Burn and Plastic Surgery, Zunyi Medical College
Other Study IDs: KLLY-2024-093
Record Dates: First submitted 2025-03-26; First posted 2025-04-10 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Gynecologic Cancer-related Lower Extremity Lymphedema; Lymphedema
MeSH Terms: conditions — Lymphedema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- VLNT + LVA + LS (Vascularized Lymph Node Transfer + Lymphaticovenular Anastomosis + Liposuction): This triple-modality intervention combines physiologic and debulking techniques. VLNT is performed to restore lymphatic function by transferring vascularized lymph nodes to the affected limb. LVA further facilitates lymphatic drainage by creating anastomoses between lymphatic vessels and nearby venules. LS is conducted to remove excess fibroadipose tissue and reduce limb volume. This comprehensive approach is hypothesized to provide synergistic and sustained benefits in severe or refractory lymphedema cases.
  Interventions: Procedure: VLNT（Vascularized Lymph Node Transfer）; Procedure: LVA（Lymphaticovenular Anastomosis）; Procedure: LS（Liposuction）
- VLNT + LS (Vascularized Lymph Node Transfer + Liposuction): This dual-modality intervention focuses on both physiologic restoration and volume reduction. VLNT is used to reconstruct lymphatic drainage pathways, while LS addresses tissue hypertrophy. This combination is selected for patients with poor lymphatic function and substantial limb volume increase, in whom LVA is not feasible due to lack of functional lymphatic vessels.
  Interventions: Procedure: VLNT（Vascularized Lymph Node Transfer）; Procedure: LS（Liposuction）
- LVA + LS (Lymphaticovenular Anastomosis + Liposuction): This approach combines a minimally invasive physiologic procedure (LVA) with LS. LVA promotes lymph flow by bypassing obstructed lymphatic channels, while LS removes accumulated fibrofatty tissue. It is suitable for patients with partially preserved lymphatic function and moderate limb volume increase.
  Interventions: Procedure: LVA（Lymphaticovenular Anastomosis）; Procedure: LS（Liposuction）

INTERVENTIONS:
Procedure: VLNT（Vascularized Lymph Node Transfer） — VLNT is a physiologic surgical procedure in which vascularized lymph nodes are harvested from a donor site (e.g., groin or submental region) and transplanted to the affected limb to restore lymphatic drainage. The transferred lymph nodes are anastomosed to recipient vessels to ensure perfusion, aiming to reconstruct lymphatic flow and reduce lymphedema-related swelling and fibrosis.
  Groups: VLNT + LS (Vascularized Lymph Node Transfer + Liposuction); VLNT + LVA + LS (Vascularized Lymph Node Transfer + Lymphaticovenular Anastomosis + Liposuction)
Procedure: LVA（Lymphaticovenular Anastomosis） — LVA is a supermicrosurgical technique designed to improve lymphatic drainage by creating anastomoses between functional lymphatic vessels and nearby venules. Under high magnification, lymphatic vessels (typically <0.8 mm) are identified and connected to subdermal venules to bypass obstructed lymphatic pathways, facilitating improved lymph flow and symptom relief in patients with early-stage lymphedema.
  Groups: LVA + LS (Lymphaticovenular Anastomosis + Liposuction); VLNT + LVA + LS (Vascularized Lymph Node Transfer + Lymphaticovenular Anastomosis + Liposuction)
Procedure: LS（Liposuction） — LS is a volume-reduction procedure used in the management of advanced lymphedema characterized by fibroadipose tissue hypertrophy. Tumescent liposuction is performed to remove excess subcutaneous adipose tissue, thereby reducing limb volume and improving limb contour. This procedure is often combined with physiologic surgical techniques for optimal long-term outcomes.

SUMMARY:
The goal of this retrospective study is to evaluate the long-term efficacy of 3L versus 2L integrated techniques in patients with gynecologic cancer-related lower extremity lymphedema (GCR-LEL). The main research question is:

Do 3L integrated techniques provide superior long-term outcomes in reducing lower extremity lymphedema compared to 2L techniques in patients with GCR-LEL?

Medical records of patients who have received either 3L or 2L integrated interventions as part of their routine clinical management for GCR-LEL were reviewed and analyzed to assess treatment outcomes over an extended follow-up period.

ELIGIBILITY:
Inclusion Criteria:

1. The patients diagnosed with gynecological cancer-related lymphedema by clinical examination are classified by the International Lymphedema Society (ISL) guidelines as Stage II to III.
2. .Aged 18-90 years.

Exclusion Criteria:

1. Lactation, for patients with pregnancy;
2. Serious heart, lung, liver, kidney disease, as well as the history of tumor patients;
3. Disease history is less than 3 months;
4. In patients with mental illness;
5. Immunodeficiency patients.

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: From January 1st of 2018 to December 31th of 2023, 125 consecutive patients with secondary lower extremity lymphedema who underwent 3L(LVA+VLNT+LS) or 2L(LVA+LS or VLNT+LS) integrated surgical treatment were identified.
Sampling Method: Non-Probability Sample
Enrollment: 125 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Change in lower limb volume (mL) measured by circumference-based calculation | Preoperative baseline vs. postoperative follow-up (e.g., 3, 6, 12 and 18 months)
  Each participant's lower limb circumference will be measured at predefined anatomical landmarks, and limb volume will be calculated using the truncated cone formula.

SECONDARY OUTCOMES:
Cellulitis Infection Rate (episodes/year) | Preoperative baseline vs. postoperative follow-up (e.g., 3, 6, 12 and 18 months)
  The incidence of cellulitis episodes per patient was assessed through retrospective chart review and clinical records. A clinically diagnosed cellulitis episode was defined by acute onset of erythema, warmth, tenderness, and edema. We compared the mean episodes per year among different surgical approach groups.
Change in Lymphoedema Quality of Life (LYMQOL) Score | Preoperative baseline vs. postoperative follow-up (e.g., 3, 6, 12 and 18 months)
  Lymphedema-specific quality of life was measured using the LYMQOL questionnaire, which includes four domains: symptoms, emotions, function, and appearance. The total LYMQOL score was calculated and compared between preoperative and postoperative assessments in different surgical groups. We evaluated both within-group (pre-to-post) and between-group differences.
Incidence of Surgical Complications | Up to 30 days post-surgery and during follow-up (e.g., 3, 6, 12 and 18 months)
  Surgical complications (e.g., flap infection, necrosis, lymphorrhea, or deep vein thrombosis) were assessed through postoperative clinical evaluations and chart review. Wound healing status was recorded, and the presence of any adverse events was documented.
Changes in Lymphoscintigraphy and Ultrasound Findings | Preoperative imaging vs. postoperative imaging at 6, 12 and 18 months
  Lymphoscintigraphy was performed to assess dermal backflow and collateral lymphatic vessel formation, while ultrasound evaluated lymph node and lymphatic vessels status (e.g., size, vascularity, viability). Postoperative changes were compared to baseline (preoperative) imaging in each group (LVA + VLNT + LS, VLNT + LS, LVA + LS).

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Burns and Plastic Surgery, Affiliated Hospital of Zunyi Medical University, Zunyi, Guizhou, China

REFERENCES:
- [Derived] Chen J, Chen Z, Wu X, Li H, Xiao S, Wei Z, Zhang Y, Deng C. Integrated surgical treatment: a new model for treating secondary extremity lymphedema based on algorithms. Front Oncol. 2026 Jan 12;15:1676803. doi: 10.3389/fonc.2025.1676803. eCollection 2025. PMID 41602404